CLINICAL TRIAL: NCT06597292
Title: Vision Improvement for Patients With Presbyopia
Brief Title: The VIS Opti-K Low Vision Aid Device Provides Vision Improvement.
Acronym: Opti-K Pres
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIS Opti-K-Presbyopia #001
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Hyperopia; Presbyopia
Keywords: Vision improvement
MeSH Terms: conditions — Hyperopia; Presbyopia

STUDY DESIGN:
Masking Description: Patient IDs will be assigned and used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Vision improvement (Experimental)
  Interventions: Device: Vision improvement

INTERVENTIONS:
Device: Vision improvement — Vision improvement for patients with refractive disorders (hyperopia and presbyopia)

SUMMARY:
The VIS Opti-K Low Vision Aid device will be used to provide vision improvement to patients with refractive disorders (hyperopia and presbyopia).

ELIGIBILITY:
Inclusion Criteria

Subjects who meet all of the following criteria are candidates for this study:

1. Male or Female
2. Any race
3. Patient is at least 40 years old.
4. Patient is pseudophakic or is phakic with no clinically significant cataract in eye(s) to be treated.
5. Patient has manifest refraction, spherical equivalent (MRSE) between -0.50 D to 2.50 D, with no more than 1.0 D of refractive cylinder, in eye(s) to be treated.
6. Patient has uncorrected distance visual acuity (UDVA) of 20/100 or better (i.e., LogMAR ≤ 0.70) in both eyes.
7. Patient has best corrected distance visual acuity (CDVA) of 20/20 or better (i.e., LogMAR ≤ 0.00) in both eyes.
8. Patient has uncorrected near visual acuity (UNVA) between 20/50 (LogMAR 0.40) and better than 20/100 (LogMAR < 0.70) in eye(s) to be treated.
9. Patient has best corrected near visual acuity (CNVA) of at least 20/20 (LogMAR ≤ 0.00) in eye(s) to be treated.
10. Patient requires reading adds of +1.0 to +3.0 D in eye(s) to be treated.
11. Patient is not a contact lens (CL) wearer.
12. Patient has normal corneal topography.
13. Patient is willing and able to comply with all examinations.
14. Patient must be competent to sign an informed consent form before study entry.

Exclusion Criteria

Subjects who meet any of the following criteria are to be excluded from this study:

1. Corneal disease or corneal disorder in either eye.
2. Any active ocular surface disease of any severity.
3. Increased IOP (above 20 mm Hg), glaucoma or history of glaucoma.
4. Previous corneal surgery in the eye to be treated.
5. Conjunctivochalasis
6. Nystagnus
7. Diabetes
8. Pregnancy
9. Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable as a candidate for study participation or that may confound the outcome of the study.

nclusion Criteria: -

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | Up to 24 months post-treatment
  Uncorrected distance visual acuity (UDVA) is to be measured and reported using standard ETDRS visual acuity charts. UDVA change from baseline is also to be reported.
Uncorrected Near Visual Acuity (UNVA) | Up to 24 months post-treatment
  Uncorrected near visual acuity (UNVA) is to be measured and reported using standard near visual acuity charts. UNVA change from baseline is also to be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berry, PhD, Study Director — VIS, Inc.
Locations (2):
- VIS, Inc., Austin, Texas, United States
- Clarity Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No